CLINICAL TRIAL: NCT06710366
Title: Prevalence of DAO (diamino Oxidase) Deficiency in Newborns
Acronym: DAO-NEO-2022
Status: Completed | Type: Observational
Sponsor: AB Biotek (Industry)
Collaborators: Grupo Hospitalario Quironsalud-Catalunya (Unknown); Hospital Universitari General de Catalunya (Other); Quironsalud (Other)
Responsible Party: Sponsor
Other Study IDs: DAO-NEO-2022
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: DAO Genetic Variants
Keywords: DAO deficiency; DAO deficiency prevalence; AOC1 gene variants; SNPs; single-nucleotide polymorphisms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Newborns: Newborns born at the centre

SUMMARY:
Observational study to estimate the prevalence of genetic DAO deficiency in the population.

DETAILED DESCRIPTION:
Diamine oxidase (DAO) is an enzyme encoded by the AOC1 gene responsible for the degradation of extracellular histamine. There are different factors that can induce a decrease in the DAO activity, with genetic origin being the main one. Currently, multiple genes have been identified SNPs that can alter the correct functioning of the DAO. The four most relevant SNPs that lead to a reduction in the enzymatic activity of DAO or a transcriptional activity decreased in this are the following: c.47C>T (rs10156191), c.995C>T (rs1049742), c.1990C>G (rs1049793) and c.-691G>T (rs2052129). Clinical studies indicate that DAO deficiency has a high prevalence in diseases such as Migraine (87%), fibromyalgia (75%) or attention deficit hyperactivity disorder (ADHD) in children (75%). However, to date no study has been conducted exploring the prevalence gene of DAO deficiency in the general population. Thus, the objective of this study is to estimate the prevalence of genetic DAO deficiency in the population.

ELIGIBILITY:
Inclusion Criteria:

* Newborns
* Both sexes
* Explicit acceptance of the parents or guardians of participation through the signature of the informed consent

Exclusion Criteria:

* None

Ages: 0 Days to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns born in Hospital Universitari Genreal de Catalunya during the period of study
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
AOC1 gene variants | In a range from day of birth up to 3 days of life
  DAO deficiency will be defined as the presence of at least one of the SNPs of the AOC1 gene described previously, with reference rs10156191, rs1049742, rs1049793 and rs2052129

SECONDARY OUTCOMES:
Sex | In a range from day of birth up to 3 days of life
  Sex
Demographic characteristics | In a range from day of birth up to 3 days of life
  Ethnicity

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
AOC1 genetic SNPs prevalence in the studied population
Supporting Information: Study Protocol, ICF, CSR
Time Frame: According to legislation

REFERENCES:
- [Background] Blasco-Fontecilla H, Bella-Fernandez M, Wang P, Martin-Moratinos M, Li C. Prevalence and Clinical Picture of Diamine Oxidase Gene Variants in Children and Adolescents with Attention Deficit Hyperactivity Disorder: A Pilot Study. J Clin Med. 2024 Mar 14;13(6):1659. doi: 10.3390/jcm13061659. PMID 38541885
- [Background] Lopez Garcia R, Ferrer-Garcia J, Sansalvador A, Quera-Salva MA. Prevalence of Diamine Oxidase Enzyme (DAO) Deficiency in Subjects with Insomnia-Related Symptoms. J Clin Med. 2024 Aug 6;13(16):4583. doi: 10.3390/jcm13164583. PMID 39200725
- [Background] Ponce Diaz-Reixa J, Aller Rodriguez M, Martinez Breijo S, Suanzes Hernandez J, Ruiz Casares E, Perucho Alcalde T, Bohorquez Cruz M, Mosquera Seoane T, Sanchez Merino JM, Freire Calvo J, Fernandez Suarez P, Chantada Abal V. Lower Urinary Tract Symptoms (LUTS) as a New Clinical Presentation of Histamine Intolerance: A Prevalence Study of Genetic Diamine Oxidase Deficiency. J Clin Med. 2023 Oct 31;12(21):6870. doi: 10.3390/jcm12216870. PMID 37959335
- [Background] Izquierdo-Casas J, Comas-Baste O, Latorre-Moratalla ML, Lorente-Gascon M, Duelo A, Vidal-Carou MC, Soler-Singla L. Low serum diamine oxidase (DAO) activity levels in patients with migraine. J Physiol Biochem. 2018 Feb;74(1):93-99. doi: 10.1007/s13105-017-0571-3. Epub 2017 Jun 17. PMID 28624934
- [Background] Schnedl WJ, Lackner S, Enko D, Schenk M, Holasek SJ, Mangge H. Evaluation of symptoms and symptom combinations in histamine intolerance. Intest Res. 2019 Jul;17(3):427-433. doi: 10.5217/ir.2018.00152. Epub 2019 Mar 7. PMID 30836736